CLINICAL TRIAL: NCT03250208
Title: Probiotics and the Female Urinary Microbiome ProFUM Trial (Probiotics Effect on the Female Urinary Microbiome)
Brief Title: Probiotics Effect on the Female Urinary Microbiome ProFUM Trial (Probiotics Effect on the Female Urinary Microbiome)
Acronym: ProFUM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Elizabeth Mueller, Associate Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 209830
Record Dates: First submitted 2017-07-19; First posted 2017-08-15 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Healthy
Keywords: Microbiome; Lactobacillus; Probiotic; Fem-Dophilus
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Participants are randomized to receive placebo or a probiotic using a 1:2 allocation, respectively
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participants and research team members are masked in this randomized placebo-controlled trial. The investigational pharmacist is unmasked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): Participants randomized to this group will take two placebo capsules daily during days 21-60.
  Interventions: Other: Placebo
- Intervention group (Experimental): The intervention in this study is a probiotic. Participants randomized to this group will take two capsules of a probiotic daily during days 21-60
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — Participants randomized to the intervention group will receive Women's Fem Dophilus ® by Jarrow Formulas.
  Other Names: Fem Dophilus
  Arms: Intervention group
Other: Placebo — Participants randomized to the control group will receive a placebo containing no active ingredients
  Other Names: Inactive substance
  Arms: Control Group

SUMMARY:
The study will enroll healthy pre-menopausal female volunteers in the community. These subjects will act as their own controls. The subjects will collect voided urine and peri-urethral swab specimens daily for several months. They will also be asked to collect vaginal and peri-rectal swab specimens at various time points. Subjects will document various lifestyle variables daily. During the middle of the study, subjects will be randomized to probiotic vs placebo. Using bacterial culture and 16S rRNA gene sequencing, the study will measure the bacterial populations of several anatomic sites longitudinally: voided urine, peri-urethra, vagina, and peri-rectal. The study hypothesizes that oral probiotic usage will alter the bacterial populations and ratio of Lactobacillus to E. coli within each of these sites. Additionally, the study hypothesizes that the changes within each site will occur first in the rectum (i.e. GI tract), followed by the vagina, and then the urethra and bladder.

Using the prospective design of daily sampling and lifestyle variable documentation, the study may be able to identify possible influences on microbiome stability within the sampled sites. The lifestyle variables recorded include: diet, medication usage, menstruation, sexual activity, and alcohol consumption.

This pilot study will establish the variance of the outcome variables among healthy women and confirm the emergence of the probiotic with the recommended dose. With this information, future researchers will be able to calculate the power needed for a larger randomized trial. This trial would also randomize patients who may be at risk for a UTI to receive a probiotic vs placebo. The primary outcome measurement will be the change in the ratio of Lactobacillus to E. coli. As a secondary aim, the study will evaluate the incidence of UTI in the patients.

DETAILED DESCRIPTION:
In this study, the primary aim is to identify the change in the Lactobacillus E. coli ratio within the lower urinary tract, the vagina, and the peri-rectal area in response to an oral probiotic as well as to evaluate the stability of these changes following cessation of an oral probiotic. Voided urine and peri-urethral, vaginal, and peri-rectal swab samples will be analyzed for their Lactobacillus E. coli ratio using bacterial culture as well as 16S ribosomal RNA gene sequencing. The study will compare the ratios present before, during, and after oral probiotic usage. The study will also compare the change in ratios between subjects taking the oral probiotic and those taking an oral placebo.

A secondary aim is to identify the normal daily changes (i.e. stability) in the bacterial populations within the voided urine, including whether host intrinsic (e.g. diet, hygiene, and sexual activity) and extrinsic (e.g. menstruation) factors affect the stability of bacterial populations. The bacterial populations defining the voided urine samples will be correlated to various daily subject-reported lifestyle variables. These include diet, hygiene, sexual activity, medication usage, alcohol usage, menstruation, and urinary-related symptoms. These lifestyle variables will be recorded each day for the entire duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal healthy women in the community (As defined by presence of menses at least once in the last 12 months).
* Age 18 years or older.
* Agreement to collect daily samples (varying combinations of voided, periurethral, and perianal swabs) for 3 months and bring the samples to Loyola University Medical Center
* Agree to record and return a daily lifestyle diary
* Understand and agree to taking daily oral probiotic or placebo while being blinded
* Able to read and speak English
* Able to obtain clean-catch urine

Exclusion Criteria:

* Non-English speaking women
* Allergy or contraindication to the probiotic used in this study
* Prior participation in the study
* Currently pregnant or lactating or planning a pregnancy within 6 months of consenting to participate in the study
* Inability to obtain a 'clean catch' urine sample
* Subjects with an indwelling catheter
* Males are excluded from participation
* Women planning time away for more than 7 days following consent to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Lactobacillus E. coli ratio in the rectum | 95 days
  We will measure participants' rectal Lactobacillus E. coli ratio at baseline and after treatment. The change in this ratio will be recorded for each participant and compared between the placebo and intervention groups.

SECONDARY OUTCOMES:
Change in Lactobacillus E. coli ratio in the vagina | 95 days
  We will measure participants' vaginal Lactobacillus E. coli ratio at baseline and after treatment. The change in this ratio will be recorded for each participant and compared between the placebo and intervention groups.
Change in Lactobacillus E. coli ratio in the urethra | 95 days
  We will measure participants' urethral Lactobacillus E. coli ratio at baseline and after treatment. The change in this ratio will be recorded for each participant and compared between the placebo and intervention groups.
Prevalence of urinary tract infections | 95 days
  At the final study visit, we will record whether each participant experienced or did not experience a urinary tract infection (UTI). The odds of a UTI among those in the intervention cohort will be compared to the odds of a UTI in the placebo cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Mueller, MD, Principal Investigator — Loyola University Health System
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available

REFERENCES:
- [Background] Urinary Incontinence Treatment Network (UITN). The Trial of Mid-Urethral Slings (TOMUS): Design and Methodology. J Appl Res. 2008;8(1):AlboVol8No1. PMID 24772006
- [Background] FitzGerald MP, Brubaker L. Colpocleisis and urinary incontinence. Am J Obstet Gynecol. 2003 Nov;189(5):1241-4. doi: 10.1067/s0002-9378(03)00642-2. PMID 14634547
- [Background] Fitzgerald MP, Richter HE, Bradley CS, Ye W, Visco AC, Cundiff GW, Zyczynski HM, Fine P, Weber AM; Pelvic Floor Disorders Network. Pelvic support, pelvic symptoms, and patient satisfaction after colpocleisis. Int Urogynecol J Pelvic Floor Dysfunct. 2008 Dec;19(12):1603-9. doi: 10.1007/s00192-008-0696-6. Epub 2008 Aug 9. PMID 18690402
- [Background] Fok CS, McKinley K, Mueller ER, Kenton K, Schreckenberger P, Wolfe A, Brubaker L. Day of surgery urine cultures identify urogynecologic patients at increased risk for postoperative urinary tract infection. J Urol. 2013 May;189(5):1721-4. doi: 10.1016/j.juro.2012.11.167. Epub 2012 Dec 3. PMID 23219547
- [Background] Foxman B, Cronenwett AE, Spino C, Berger MB, Morgan DM. Cranberry juice capsules and urinary tract infection after surgery: results of a randomized trial. Am J Obstet Gynecol. 2015 Aug;213(2):194.e1-8. doi: 10.1016/j.ajog.2015.04.003. Epub 2015 Apr 13. PMID 25882919
- [Background] Beerepoot MA, ter Riet G, Verbon A, Nys S, de Reijke TM, Geerlings SE. [Non-antibiotic prophylaxis for recurrent urinary-tract infections]. Ned Tijdschr Geneeskd. 2006 Mar 11;150(10):541-4. Dutch. PMID 16566416
- [Background] Wilton L, Kollarova M, Heeley E, Shakir S. Relative risk of vaginal candidiasis after use of antibiotics compared with antidepressants in women: postmarketing surveillance data in England. Drug Saf. 2003;26(8):589-97. doi: 10.2165/00002018-200326080-00005. PMID 12825971
- [Background] Hooton TM. Recurrent urinary tract infection in women. Int J Antimicrob Agents. 2001 Apr;17(4):259-68. doi: 10.1016/s0924-8579(00)00350-2. PMID 11295405
- [Background] Raz R, Stamm WE. A controlled trial of intravaginal estriol in postmenopausal women with recurrent urinary tract infections. N Engl J Med. 1993 Sep 9;329(11):753-6. doi: 10.1056/NEJM199309093291102. PMID 8350884